CLINICAL TRIAL: NCT01946386
Title: A Vasoconstriction Study With LEO 90100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LP0053-69
Record Dates: First submitted 2013-09-11; First posted 2013-09-19 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-07

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 90100 (Experimental)
  Interventions: Drug: LEO 90100 Aerosol, foam; Drug: Betamethasone dipropionate in LEO 90100 Aerosol, foam, vehicle; Drug: LEO 90100 Aerosol, foam, vehicle; Drug: Daivobet® ointment; Drug: Dermovate® cream; Drug: Synalar® ointment

INTERVENTIONS:
Drug: LEO 90100 Aerosol, foam — The products will be applied on 6 test sites (according to random assignment to specific test sites predetermined on their anterior face of forearms) for 6 hours
Drug: Betamethasone dipropionate in LEO 90100 Aerosol, foam, vehicle
Drug: LEO 90100 Aerosol, foam, vehicle
Drug: Daivobet® ointment
Drug: Dermovate® cream
Drug: Synalar® ointment

SUMMARY:
The purpose of this study is to compare the pharmacodynamic activity of LEO 90100 with Dermovate® cream, Dovobet® ointment, betamethasone dipropionate in LEO90100 vehicle, Synalar® ointment and LEO 90100 vehicle using a human skin blanching test.

ELIGIBILITY:
Inclusion Criteria:

* Following verbal and written information about the trial, the subject must provide signed and dated informed consent before any study related activities are carried out.
* Healthy male or female volunteers, 18 to 50 years old, both inclusive

Exclusion Criteria:

* Female subjects who are pregnant or who are breast feeding.
* Abnormal pigmentation of the skin or skin type that could, in any way, confound interpretation of the study results (skin type V and VI on the Fitzpatrick scale)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Visual assessment of skin blanching (visual score (VS)) | 06:10, 08:00, 10:00, 12:00, 24:00, 28:00 and 32:00 hours after application
  Visual Assessment of Skin Blanching on scores 0 to 4

SECONDARY OUTCOMES:
Change from baseline in colorimetric parameter a* (the red/green balance) at each time point | 06:10, 08:00, 10:00, 12:00, 24:00, 28:00 and 32:00 hours after application
  Change from baseline in colorimetric parameter. AUC (0-32h) of this change by treatment site will be calculated after subtraction of untreated site change
Change from baseline in colorimetric parameter L* (luminance) at each time point (ΔL*) | 06:10, 08:00, 10:00, 12:00, 24:00, 28:00 and 32:00 hours after application
  AUC (0-32h) of this change by treatment site will be calculated after subtraction of untreated site change

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- CPCAD, Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Queille-Roussel C, Bang B, Clonier F, Lacour JP. Phase I evaluation of the vasoconstrictor potential of an innovative fixed combination calcipotriene plus betamethasone dipropionate aerosol foam versus other corticosteroid psoriasis treatments. J Am Acad Dermatol. 2015:72 Suppl 1;AB243 (P915).
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en